CLINICAL TRIAL: NCT02079883
Title: Ocriplasmin Research to Better Inform Treatment (ORBIT)
Acronym: ORBIT
Status: Completed | Type: Observational
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Other Study IDs: TG-MV-018
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Symptomatic Vitreomacular Adhesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — No biospecimens collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ocriplasmin

SUMMARY:
This is a multicenter, prospective, observational, Phase 4 study that will assess clinical outcomes and safety of JETREA® administered in a real-world setting for the treatment of symptomatic vitreomacular adhesion (VMA) by assessing anatomical and functional outcomes in 1500 patients recruited across approximately 120 USA retina sites.

DETAILED DESCRIPTION:
The sites will prospectively enroll consecutive patients eligible for participation in the study. Informed consent will be obtained prior to any data being collected. This study is observational; therefore, all treatment decisions and assessments are at the discretion of the patient's treating physician and are not mandated by the study design or protocol. Patients will be enrolled at a routinely scheduled visit, on the day of JETREA® administration after the JETREA® injection. No specific visits, examinations, laboratory tests or procedures are mandated as part of this study. There is no pre-set visit schedule, and the frequency and timing of actual patient visits is at the discretion of the treating physician following standard of care. All available and relevant data will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older diagnosed with symptomatic VMA treated with JETREA ® at the physician's discretion in a manner consistent with the product label.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients who are treated with JETREA® for medical conditions outside of the US product label.
* Concurrent participation in a research study that prescribes ocular treatment, imaging and/or interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will assess clinical outcomes and safety in patients treated with JETREA® administered in a real-world setting for the treatment of symptomatic VMA
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Resolution of VMA by Spectral-domain optical coherence tomography (SD-OCT) as determined by the treating physician. | 12 Months
Full thickness macular hole (FTMH) closure by SD-OCT as determined by the treating physician | 12 months
Mean change in visual acuity (VA) from baseline across time | 12 months
Occurrence and time to vitrectomy | 12 months

OTHER OUTCOMES:
Monitoring of adverse drug reactions (ADRs) | 12 months
Change from baseline in ocular signs and symptoms across time. | 12 months

CONTACTS AND LOCATIONS:
Locations (110):
- United States (110):
  - Retinal COnsultants of Arizona, Phoenix, Arizona
  - Associated Retina Consultants, Ltd, Phoenix, Arizona
  - Retina Vitreous Assciates Medical Group, Beverly Hills, California
  - Valley Retina Institute, PA, Encino, California
  - California Eye Institute, Fresno, California
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Retina Associates of Orange County, Laguna Hills, California
  - South Coast Retina Center, Long Beach, California
  - University of Southern California Medical Center, Los Angeles, California
  - Jules Stein Eye Institute, Los Angeles, California
  - University of California at Irvine Medical Center, Orange, California
  - Southern California Desert Retina Specialists, Palm Springs, California
  - Lawrence J. Ellison Ambulatory Care Center - UC Health, Sacramento, California
  - Retinal Diagnostic Center, San Jose, California
  - Orange County Retina Medical, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Colorado Retina Associates, Golden, Colorado
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Retina Macula Specialists of Miami, Miami, Florida
  - MedEye Associates, Miami, Florida
  - Bascom-Palmer, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Center for Sight, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Vitreous Associates of FL, St. Petersburg, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, Decatur, Georgia
  - Marietta Eye, Marietta, Georgia
  - Retina Consultants of Hawaii, Inc, ‘Aiea, Hawaii
  - Chicagoland Retinal Consultants, Chicago, Illinois
  - Lions of Illinois Research Institute-Eye and Ear Infirmary, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Retina and Macula Associates, P.C., Oak Forest, Illinois
  - Illinois Retina Center, Springfield, Illinois
  - Carle Research Institute, Urbana, Illinois
  - Dr. Thomas Ciulla, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Sabates Eye Centers, Leawood, Kansas
  - Vitreo-Retinal Consultants & Surgeons, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Eye Specialists of Louisville, PSC, Louisville, Kentucky
  - Carl W Baker, Paducah, Kentucky
  - Retina & Vitreous of Louisiana, Baton Rouge, Louisiana
  - Acadiana Retina Consultants, Lafayette, Louisiana
  - Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, PA, Baltimore, Maryland
  - The Retina Group of Washintong, Chevy Chase, Maryland
  - Katzen Eye Group, Lutherville, Maryland
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Vitroretinal Assciates, Worcerster, Massachusetts
  - Central Mass Retina & Uveitis Center, Worcester, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Vitreo Retinal Surgery, Minneapolis, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - niversity of Nebraska Medical Center, Omaha, Nebraska
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Eyesight Ophthalmic Services, Portsmouth, New Hampshire
  - Retina Center of New Jersey, LLP, Bloomfield, New Jersey
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - NJ Retina, New Brunswick, New Jersey
  - Retinal and Ophthalmic Consultants, Northfield, New Jersey
  - Retina Associates Of New Jersey, Pa, Teaneck, New Jersey
  - Kwiat Eye & Laser Surgery, Amsterdam, New York
  - Capital Retina Associates, Latham, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - MaculaCare, New York, New York
  - Vitreous-Retina-Macula Consultants of NY,PC, New York, New York
  - Island Retina, Shirley, New York
  - Retina Vitreous Surgeons of Central NY, Syracuse, New York
  - Capital Region Retina, Wilton, New York
  - Duke University Eye Center, Durham, North Carolina
  - East Carolina Retina Consultants, Greenville, North Carolina
  - North Carolina Retina Assoc, Raleigh, North Carolina
  - Cape Fear Retina, Wilmington, North Carolina
  - Dr Mark Nelson, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Tri-State Centers for Sight, Cincinnati, Ohio
  - Eye Care Associates of Greater Cincinnati, Inc., Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Retina Associates of Cleveland, Middleburg Heights, Ohio
  - Retina Vitreous Center in Edmond Oklahoma, Edmond, Oklahoma
  - Pennsylvania Retina Specialists PC, Camp Hill, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Associates Ophthalmology and Associates Surgery Centers, LLC, Pittsburgh, Pennsylvania
  - Allegheny Ophthalmology and Orbital Associates, Pittsburgh, Pennsylvania
  - Carolina Eyecare, Charlestown, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, Kingsport, Tennessee
  - Eye Health Partners & Vision America, Nashville, Tennessee
  - Retina Research Center, Austin, Texas
  - Texoma Retina Center, Denison, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retina Specialists, Plano, Texas
  - Medical Center Ophthamalogy Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Eye Care Associates, Tyler, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - The Retina Group of Washington, Fairfax, Virginia
  - Wagner Macula and Retina Center, Virginia Beach, Virginia
  - Northwest Eye Surgeons, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Khanani AM, Duker JS, Heier JS, Kaiser PK, Joondeph BC, Kozma P, Rosberger DF, MacCumber M, Boyer DS, Pieramici DJ. Ocriplasmin Treatment Leads to Symptomatic Vitreomacular Adhesion/Vitreomacular Traction Resolution in the Real-World Setting: The Phase IV ORBIT Study. Ophthalmol Retina. 2019 Jan;3(1):32-41. doi: 10.1016/j.oret.2018.07.011. Epub 2018 Jul 25. PMID 30935657